CLINICAL TRIAL: NCT00860795
Title: Study of the Immunologic Effects of Echinacea Purpurea in Adults
Brief Title: Immunologic Effects of Echinacea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, James Taylor, School of Medicine: Pediatrics, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 09A1236; 5U01AT002400 (NIH)
Record Dates: First submitted 2009-03-10; First posted 2009-03-12 (Estimated); Results first posted 2010-11-17 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Upper Respiratory Tract Infections
Keywords: Echinacea; prevention; immune modulation
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Echinacea extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Echinacea (Active Comparator)
  Interventions: Biological: Echinacea purpurea
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Biological: Echinacea purpurea — Echinacea purpurea 100 mg/ml, 25 ml daily in 2 divided doses for 10 days
  Arms: Echinacea
Drug: placebo — placebo 25 ml daily in 2 divided doses for 10 days
  Arms: placebo

SUMMARY:
The goal of this study is to determine if Echinacea purpurea stimulates the immune system. For the study, 20 healthy adults will be randomized to receive Echinacea purpurea or placebo for 10 days. Blood will be drawn to assess immune markers just before beginning the study medication, during the 10 day course of medication and after completing the course of medication. It is postulated that adults receiving the Echinacea will have evidence of immune stimulation and those receiving placebo will not.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 21-65 years old
* If female of child-bearing potential, willing to use contraception to prevent pregnancy
* Speaks and reads English
* No use of any medication (other than multivitamins, essential fatty acids or probiotics)
* Willing to abstain from ingesting edible mushrooms throughout study
* Willing to eat less than 2 garlic cloves per day throughout study

Exclusion Criteria:

* Positive pregnancy test or currently breastfeeding
* History of autoimmune disease
* History of allergic rhinitis
* History of physician diagnosed eczema
* Known allergic reaction to Echinacea or related species, specifically ragweed (Ambrosia), chamomile (Matricaria), goldenrod (Solidago) and sunflower (Helianthus)
* Use of any medication within 30 days prior to first dose of study medication that is a known inhibitor or inducer of CYP34A

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-03; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A Taylor, MD, Principal Investigator — University of Washington
Locations (1):
- Bastyr University, Kenmore, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adults were recruited using general advertising and enrolled between March and August 2009
Groups:
- Echinacea; Placebo: 25 ml daily in 2 divided doses for 10 days
Period: Overall Study
Arm/Group | Echinacea | Placebo
Started | 10 | 10
Number to Complete Study Medication | 9 | 10
Completed | 10 (One participant discontinued study medication on day 5, but completed safety evaluations) | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Echinacea | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (12.6) | 37.4 (14.3) | 36.5 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Maximal Level of Tumor Necrosis Factor Alpha (pg/ml)
Description: tumor necrosis factor alpha NK cells and evidence of CD25/69 activation
Time Frame: 10 days
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: tumor necrosis alpha level (pg/ml)
Arm/Group | Echinacea | Placebo
Number analyzed (Participants) | 10 | 10
tumor necrosis alpha level (pg/ml) | 2694 (1299) | 2648 (1625)
Statistical Analysis 1: Comparison: Echinacea vs Placebo; Test type: Superiority or Other; p = .17, Regression, Linear

2. Secondary Outcome: Maximal Levels of Interferon Alpha (pg/ml)
Description: interferon alpha was measured on days 2, 3, 7, 10 in peripheral blood mononuclear cells. The highest level on any of these days in each participant was chosen as the maximal level and used for the analysis.
Time Frame: 10 days
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: interferon alpha level (pg/ml)
Arm/Group | Echinacea | Placebo
Number analyzed (Participants) | 10 | 10
interferon alpha level (pg/ml) | 29 (47) | 35 (69)
Statistical Analysis 1: Comparison: Echinacea vs Placebo; Test type: Superiority or Other; p = .72, Regression, Linear

3. Secondary Outcome: Maximal CD25/69 Activation (% of NK CD25/69+ Cells)
Description: NK cells with evidence of CD25/69 activation were assessed on days 2, 3, 7, and 10. The highest percentage found on one of these days in each participant was categorized as the the maximal CD25/69 activation
Time Frame: 10 days
Population: intention to treat
Measure: Mean (Standard Deviation); unit: (% of NK CD25/69+ cells)
Arm/Group | Echinacea | Placebo
Number analyzed (Participants) | 10 | 10
(% of NK CD25/69+ cells) | 1.07 (.70) | 1.53 (1.10)
Statistical Analysis 1: Comparison: Echinacea vs Placebo; Test type: Superiority or Other; p = .2, Regression, Linear

4. Secondary Outcome: Adverse Effects
Time Frame: 30 days
Population: intention to treat
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Echinacea | Placebo
Number analyzed (Participants) | 10 | 10
participants
  constipation | 1 | 1
  blurred vision | 1 | 1
  diarrhea | 0 | 1
  gas/indigestion | 1 | 2
  nausea | 4 | 1
  taste: abnormal/metallic | 1 | 1
  musculoskeletal pain | 0 | 1
  headache | 0 | 3
  fever | 1 | 0
  sore throat | 0 | 1
  nasal congestion | 1 | 1
  rash | 1 | 1
  anxiety | 1 | 2
  insomnia | 0 | 1
  weakness/fatigue | 1 | 1
  urinary: difficult/painful | 0 | 1
  other | 4 | 2

5. Secondary Outcome: Maximal Levels of Interleukin 2 (pg/ml)
Description: interleukin 2 was measured on days 2, 3, 7, 10 in peripheral blood mononuclear cells. The highest level on any of these days in each participant was chosen as the maximal level and used for the analysis.
Time Frame: 10 days
Population: intention to treat
Measure: Mean (Standard Deviation); unit: interleukin 2 level (pg/ml)
Arm/Group | Echinacea | Placebo
Number analyzed (Participants) | 10 | 10
interleukin 2 level (pg/ml) | 287 (244) | 829 (1072)
Statistical Analysis 1: Comparison: Echinacea vs Placebo; Test type: Superiority or Other; p = .51, Regression, Linear

6. Secondary Outcome: Maximal Levels of Interleukin 6 (pg/ml)
Description: interleukin 6 was measured on days 2, 3, 7, 10 in peripheral blood mononuclear cells. The highest level on any of these days in each participant was chosen as the maximal level and used for the analysis.
Time Frame: 10 days
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: interleukin 6 level (pg/ml)
Arm/Group | Echinacea | Placebo
Number analyzed (Participants) | 10 | 10
interleukin 6 level (pg/ml) | 5085 (375) | 2862 (8761)
Statistical Analysis 1: Comparison: Echinacea vs Placebo; Test type: Superiority or Other; p = .43, Regression, Linear

7. Secondary Outcome: Maximal Levels of Interleukin 12 (pg/ml)
Description: interleukin 12 was measured on days 2, 3, 7, 10 in peripheral blood mononuclear cells. The highest level on any of these days in each participant was chosen as the maximal level and used for the analysis.
Time Frame: 10 days
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: interleukin 12 level (pg/ml)
Arm/Group | Echinacea | Placebo
Number analyzed (Participants) | 10 | 10
interleukin 12 level (pg/ml) | 13 (17) | 6 (19)
Statistical Analysis 1: Comparison: Echinacea vs Placebo; Test type: Superiority or Other; p = .61, Regression, Linear

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Echinacea | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 6/10 | 7/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Echinacea (N=10) | Placebo (N=10)
blurred vision (Eye disorders) | 1 | 0
constipation (Gastrointestinal disorders) | 1 | 1
diarrhea (Gastrointestinal disorders) | 0 | 1
gas/indigestion (Gastrointestinal disorders) | 1 | 2
nausea (Gastrointestinal disorders) | 4 | 1
taste: abnormal/metallic (Gastrointestinal disorders) | 1 | 1
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
headache (General disorders) | 0 | 3
urinary: difficult/painful (Renal and urinary disorders) | 0 | 1
fever (General disorders) | 1 | 0
sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
rash (Skin and subcutaneous tissue disorders) | 1 | 1
anxiety (Nervous system disorders) | 1 | 2
insomnia (General disorders) | 0 | 1
weakness/fatigue (General disorders) | 1 | 1
other (General disorders) | 4 | 2 — tongue tingling, tongue numbness, lip numbness reported by 3 participants taking Echinacea

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No